CLINICAL TRIAL: NCT05190549
Title: CAV Regimen (Cladribine Combined With Low Dose Ara-C and Venetoclax) Pretreatment Followed by Hematopoietic Stem Cell Transplantation for Relapsed or Refractory Acute Leukemia: a Multi-center, Open-label and Prospective Clinical Trial
Brief Title: CAV Regimen Bridging to HSCT for R/R AL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The Second People's Hospital of Huai'an (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Prof., The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZRRAL01
Record Dates: First submitted 2022-01-04; First posted 2022-01-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Acute Leukemia, Relapsed; Acute Leukemia Refractory
Keywords: CAV regimen; HSCT
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAV Regimen Bridging to HSCT (Experimental)
  Interventions: Procedure: CAV regimen bridging to HSCT

INTERVENTIONS:
Procedure: CAV regimen bridging to HSCT — The enrolled patients will be firstly given CAV bridging regimen (cladribine 5mg/m2/ day for 5 days, cytarabine 20mg q12h for 10 days, and began at 100 mg on day 1 and increased stepwise over 3 days to reach the target dose of 400 mg (100 mg, 200 mg, and 400 mg) on days 1-21. Conditioning regimen for allo-HSCT may be administrated after completion of the CAV regimen, with or without consolidation therapy.

SUMMARY:
Although allogeneic hematopoietic stem cell transplantation (HSCT) is a curative treatment option for acute leukemia (AL), relapsed or refractory (R/R) AL is still a big challenge. It is believed that decreased tumor burden before HSCT is a favorable factor contributing to the long-term survival of R/R AL patients and many kinds of bridging chemotherapy regimens were devised to kill leukemic cells before HSCT, there is still no consensus that which regimen is optimal. This study is to investigate the curative efficacy and safety of bridging CAV (cladribine combined with low dose Ara-C and venetoclax) regimens followed by HSCT treatment protocol for R/R AML.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AL must meet one of the following criteria ：A or B. A: relapsed AL disease was defined as follows: (1) Reappearance of leukemic blasts in the peripheral blood after CR; or (2) detection of >5% blasts in the bone marrow (BM) not attributable to another cause(e.g. regeneration after consolidation therapy); or (3) extramedullary relapse.

   B: refractory AL disease was defined as follows: (1) failure to achieve CR, CRh or CRi after two courses of intensive induction treatment. or (2) failure to achieve complete remission after one cycle of induction chemotherapy or a reduction in the number of blasts of less than 50% after one cycle of induction treatment, with residual blasts >15%.
2. patients without ≥grade 3 of cardiac, hepatic, pulmonary, or renal dysfunctions.
3. sign informed consent voluntarily.
4. Patients aged between 16 and 70 years old, male or female is permitted.
5. ECOG performance status score less than 1.
6. The expected survival is longer than 3 months.

Exclusion Criteria:

1. With other malignant tumors.
2. Patients received the treatment of cladribine or venetoclax.
3. Patients received cardiac angioplasty or stent implantation.
4. Active infections that are not under clinical control (bacteria or fungus or virus is included).
5. Liver functions abnormalities (total bilirubin>1.5 times the upper limit of the normal range, ALT/AST>2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST>1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine>1.5 times the upper limit of normal value).
6. Pregnant or nursing women.
7. Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met.
8. Patients participated in any other clinical trials 3 months prior to signing the informed consent.
9. Patients not suitable for the study according to the investigator's assessment.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-11-17 (Actual)

PRIMARY OUTCOMES:
ORR (overall response rate) | 1 month
  ORR was calculated as the sum of CR, CRi, MLFS and PR.

SECONDARY OUTCOMES:
OS (Overall survival) | 1 year
  OS was defined as the time from enrollment to this study to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
EFS (Event-free survival) | 1 year
  EFS was defined as the time from the initiation of CAV to treatment failure, relapse, death from any cause or the last follow-up.
Adverse events (AEs) | 2 months
  It is evaluated and graded according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Li Xue, M.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes